CLINICAL TRIAL: NCT03879200
Title: Group Antenatal Care for Somali Born Women: a Feasibility Study Including Intervention Development and Evaluation
Brief Title: Group Antenatal Care for Somali Born Women
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Limited time frame and financial resources. The anticipated increase of eligable migrant women did not occur during the period because of changes in migration policies.
Sponsor: Karolinska Institutet (Other)
Collaborators: Uppsala University (Other); La Trobe University (Other); Dalarna University (Other)
Responsible Party: Principal Investigator, Erica Schytt, Associate professor, Karolinska Institutet
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Prevention
Other Study IDs: Group Antenatal Care, Somali
Record Dates: First submitted 2016-09-28; First posted 2019-03-18 (Actual); Last update posted 2020-11-03 (Actual); Status verified 2020-10

CONDITIONS: Antenatal Care; Immigrant; Pregnancy

STUDY DESIGN:
Intervention Model Description: Recruitment of controls conducted meanwhile developing the intervention in collaborations with Somali born women, partners, midwives and project steering group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard Individual care (No Intervention): Historical controls Individual care follows standard individual Swedish antenatal care, i.e.8-9 30 minutes appointments with a midwife during a normal pregnancy including information and regular pregnancy check-ups. Women are offered classes (3 x 2 hours) that provide preparation for birth and parenthood according to the same guidelines. Obstetricians and general practitioners have a consultant role.
- Group antenatal care (Experimental): Group antenatal care will follow the same guidelines as for individual care but with tailored content provided in language supported group sessions.
  Interventions: Other: Group antenatal care

INTERVENTIONS:
Other: Group antenatal care — Care will be provided in group sessions in dialogue sensitive to language and cultural issues. Group numbers will be around 8; the woman with partner or other companion welcome. The content of the sessions will be designed in collaboration with midwives and Somali born women, following the present parental education and findings from the focus groups. The sessions will be held at the antenatal clinic led by one or two midwife, assisted by the trained female Somali interpreter.
  Arms: Group antenatal care

SUMMARY:
Somali-born women comprise one of the largest groups of immigrant women of childbearing age in Sweden, with increased risks for perinatal morbidity and mortality and poor experiences of care. Midwives in antenatal care have expressed a need for development of care tailored for this group of women.

The overall aim is to develop and test the acceptability and immediate impacts of group antenatal care for Somali women residing in Sweden, in an effort to improve their experiences of antenatal care, their knowledge about childbearing and the Swedish health care system, their emotional wellbeing and ultimately, their pregnancy outcomes.

The study includes four steps:

Step I is the preparation phase including needs assessment. Step II is the intervention development and evaluation tool development phase. Step III is the intervention phase, which includes the implementation and evaluation of the intervention using historical controls.

Step IV is the process evaluation and "lessons learned". Historical controls (n=80) have received standard individual care according to the national Swedish program for antenatal care, i.e. 8-9 appointments with a midwife during a normal pregnancy. Women in the intervention group (n=80) receive Group Antenatal Care provided in group sessions in a dialogue sensitive to language and cultural issues. The sessions are led by a midwife, assisted by a trained female Somali interpreter. 15 minutes for individual checkups in privacy are provided at end of the session.

Primary outcomes: Women's overall ratings of antenatal care and views about specific aspects of care are captured by core questions in the Migrant Friendly Maternity Care Questionnaire (MFMCQ); and emotional wellbeing by the Edinburgh Postnatal Depression Scale (EPDS).

Data are collected at recruitment, in gestational week 36 and at 2 months postpartum by means of face-to face interviews or interviews by telephone by a trained bilingual research assistant.

DETAILED DESCRIPTION:
Group antenatal care is developed in collaboration with Somali women, midwives and a reference group; to suit Somali born women's needs. The intervention is now evaluated for feasibility, acceptability and sustainability, by means of a historically controlled trial. The study is a non-randomized feasibility study in which the intervention and material has been developed parallel to the data collection for the control group; i.e. the historical controls receiving standard care.

Specific objectives for the study are;

1. To establish with Somali-born women and antenatal caregivers the acceptability and feasibility of group antenatal care and to develop an appropriate model in order to improve outcomes for Somali-born women;
2. To establish appropriate recruitment and data collection procedures and outcome measures in consultation with the Somali community and with care providers in order to evaluate the new model; and
3. To implement and evaluate an agreed model of group antenatal care in partnership with the Somali community and antenatal caregivers.

Methods:

Step I was the preparation phase, including needs assessment, the development of contextual understanding and building a logic model for the project. A project steering group comprised of research team members, antenatal care midwives and representatives of the Somali community in Borlänge and North Stockholm was formed, to inform the intervention and the study. Somali born women in local community settings were encountered to develop a fuller understanding of issues and concerns about pregnancy and birth in a new country. The idea of group antenatal care was also discussed with women antenatal care midwives for its relevance, attractiveness and feasibility, and further how to best evaluate such a model. Focus group discussions were conducted with the following groups: 1) Somali born mothers 2) Somali born fathers; all with recent birth giving experience in Sweden, and 3) antenatal care midwives in multi-cultural settings in Sweden. The discussions were tape recorded and analysed by means of thematic analyses.

Step II was the intervention development and evaluation tool development phase. The knowledge gained in the first step, was used to develop an appropriate Group Antenatal Care model in dialogue with the project steering group and midwives. The participating midwives participated in a two days education about group antenatal care facilitation of group discussions, with input from the Steering Group representatives and findings in the focus groups discussions to enhance their understanding. Participating interpreters were oriented in the Swedish antenatal care system and the concept of group antenatal care. During this phase information material regarding the study and the intervention, a manual for midwives and tools for data collection were developed, and data collection for the historical controls receiving standard care commenced.

Step III is the intervention phase, which has commenced. In this phase the implementation and evaluation of the intervention is taking place.

The intervention and intervention group: Group antenatal care

The intervention is a developed group antenatal care to suit Somali women. Group antenatal care follows the same guidelines as for individual care but with content tailored according to findings in phase 1; i.e. based on person centred principles and dialogue by the use of motivational interviewing in group. The main-part of the care is provided in group sessions in a dialogue sensitive to language and cultural issues. Group numbers are around 8; the woman and if she wishes, her partner and/or other chosen companion. The sessions is led by a midwife, assisted by the trained female Somali interpreter/advocate. Two midwives takes turns leading the sessions for continuity and back-up. Sessions will be held in the antenatal clinic. Information and discussions include for instance sharing of information about being pregnant and giving birth in Somalia and Sweden, differences in health care, role of and trust in midwives and doctors, complications during pregnancy, labour and birth, and healthy diet during pregnancy. One hour will be allocated for individual meetings with one of the midwives (the same every time) in the clinic while the group members can chat and socialise. The midwife will document attendance and compile a summary of the discussions in a checklist.

Primary outcomes: Women's overall rating of antenatal care and views about specific aspects of care are captured by a core question in the Migrant Friendly Maternity Care Questionnaire (MFMCQ) developed by the Reproductive Outcomes And Migration international research collaboration (team members Small and Essen involved), now also translated and culturally validated in Somali (by Essen) and available for use in this study. Women's emotional wellbeing is measured by the EPDS, available in a Somali translation, but not yet fully validated requiring further cultural validation as part of the development work for this study.

Secondary outcomes: Adequate number of visits are measured by the The Adequacy of Prenatal Care Utilization Index (APCUI), i.e. expected number of visits in relation to actual number adjusted for gestational week at booking visit and delivery). Social support during pregnancy, worries about the upcoming birth and knowledge about different aspects of maternity care are assessed in interviews with women. Information about birth events and infant health will be retrieved from patient records.

Data collection: The baseline measurement is conducted at recruitment, around gestational week 20. A research assistant contacts women for a face-to-face interview in a place of their choice. The interview follows the first questionnaire (Q1) including questions on background (education, occupation), migration (time in country, reason for migration, migration status, language) and social support, knowledge of the health system, pregnancy and birth and expectations about the up-coming birth.

Follow-up interviews will take place around gestational week 36 and at two months postpartum using a second and third questionnaire (Q2, Q3) with questions from the MFMCQ about experiences of care received during the pregnancy and birth and attendance at parent education classes. Maternal and infant data will be retrieved from the patient record and include the following: gestational age at the first visit, Hemoglobin, S-Ferritin, weight gain, relevant health conditions, total number of antenatal care visits, attendance at parent education, mode of birth, interventions (induction of labour, pain relief including epidural, oxytocin), blood loss, diagnoses (mother) and gestational age, birth weight, small for gestational age, large for gestational age, head circumference, Apgar score, umbilical cord pH, and the need for neonatal intensive care (infant). Midwives' experiences of different aspects of the intervention will be collected by means of individual interviews.

Control group: Historical controls: Individual care

Individual care follow the present model of care according to the national Swedish program for antenatal care, i.e.8-9 appointments with a midwife during a normal pregnancy. The visits are scheduled for 30 minutes and include information and regular pregnancy check-ups. Women are offered classes that provide preparation for birth and parenthood according to the same guidelines and the present routine at the clinic. Midwives are the primary caregivers and they meet the same women throughout pregnancy. Obstetricians and general practitioners will have a consultant role.

Recruitment for both intervention and control groups:

In line with the actual birth rates and recruitment of one third of the Somali women at both sites, 80 women have been recruited as historical controls (2017-2018) and 80 will participate in the new model (2018-2019). Inclusion criteria are Somali born women 18 years of age or beyond, both nulliparous and multiparous, <25 gestational weeks giving consent to access their patient record data. The only exclusion criterion is severe medical problem(s) requiring individual care only, as determined by the participating clinical practice.Women are invited to participate with the help of bilingual research assistants and receive verbal and written information in Somali about the study. A small gift will be offered for their baby in appreciation for taking part.

Analyses:

Differences will be described as odds ratios and 95% confidence intervals after estimation by means of logistic regression analyses. Comparison of means will be undertaken using t-tests where data are normally distributed, or medians compared using Mann-Whitney U tests if not.

Step IV consists of a process evaluation using a mixed methods approach with data collection conducted throughout the study. The process evaluation will address whether the intervention was carried out according to plan, what was achieved, if and what adaptations were needed, who was reached by the intervention, any unexpected events and to understand the mechanisms of impact and what mediated these mechanisms. The process evaluation will also address contextual factors.

ELIGIBILITY:
Inclusion Criteria:

Somali born women, both nulliparous and multiparous, <23 gestational weeks giving consent to access their patient record data

Exclusion Criteria:

Severe medical problem(s) requiring individual care only, as determined by the participating clinical practice

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 136 (Actual)
Dates: Start 2018-05-25 (Actual); Primary Completion 2020-05-16 (Actual); Study Completion 2020-05-30 (Actual)

PRIMARY OUTCOMES:
Women's overall rating of antenatal care | 2 months postpartum
  In general, were you happy with the healthcare you received? Always vs Often, Sometimes, Seldom, Never
Women's emotional wellbeing | 2 months postpartum
  Edinburgh Postnatal Depression Scale . 10-item scale. Depressive symptoms cut-off 11/12, according to validation in Swedish women. Not yet validated in Somali migrant women in Sweden.
Women's emotional wellbeing | Late pregnancy and 2 months postpartum
  Edinburgh Postnatal Depression Scale, mean values

SECONDARY OUTCOMES:
Number of visits | patient records. Just before the birth
  The Adequacy of Prenatal Care Utilization Index (APCUI)
Social support | 2 months postpartum
  sum of 6 items (inspired by the Pregnancy Risk Assessment Monitoring System (PRAMS))
Social support | Gestational week 36
  sum of 7 items (inspired by the PRAMS)
Worries about the upcoming birth | Gestational week 36
  Cambridge Worry Scale. Single item questions (not a summated rating scale). Not worried, a little worried, very worried
Anemia during pregnancy | Gestational week 36
  Patient record data: yes/no
Induction of labour | Before active phase
  Patient record data: Induction (yes/no)
Mode of birth | At birth
  Patient record data: Mode of birth: normal vaginal, instrumental vaginal, elective caesarean, emergency caesarean
Epidural analgesia for labour pain | During active phase of labour
  Patient record data: yes/no
Apgar score <7 | At 5 minutes after the birth
  Patient record data
Need for neonatal infant intensive care (NICU) | within 7 days from birth
  Patient record data: yes/no

CONTACTS AND LOCATIONS:
Overall Officials: Erica Schytt, Professor, Principal Investigator — Karolinska Institute/Centre for Clinical Research Dalarna/West Norway University
Locations (2):
- Sweden (2):
  - The Antenatal Clinic, Domnarvet, Borlänge
  - The Antenatal Care Clinic, Spånga-Tensta, Stockholm

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ahrne M, Byrskog U, Essen B, Andersson E, Small R, Schytt E. Group antenatal care compared with standard antenatal care for Somali-Swedish women: a historically controlled evaluation of the Hooyo Project. BMJ Open. 2023 Jan 25;13(1):e066000. doi: 10.1136/bmjopen-2022-066000. PMID 36697050
- [Derived] Ahrne M, Byrskog U, Essen B, Andersson E, Small R, Schytt E. Group antenatal care (gANC) for Somali-speaking women in Sweden - a process evaluation. BMC Pregnancy Childbirth. 2022 Sep 21;22(1):721. doi: 10.1186/s12884-022-05044-9. PMID 36131237
- See also: Website for the project — https://ki.se/kbh/modrahalsovard-for-utlandsfodda-kvinnor-hooyo-projektet